CLINICAL TRIAL: NCT04945447
Title: Effects of a Pharmacist Intervention in the Primary Sector on Patients Medication and Health-related Quality of Life: A Randomised Controlled Trial
Brief Title: Improving Medication Reviews to Polypharmacy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Collaborators: The Quality Unit for General Practice North Denmark Region (Unknown)
Responsible Party: Principal Investigator, Josefine Mikkelsen, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Aalborg University
Record Dates: First submitted 2021-06-09; First posted 2021-06-30 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Polypharmacy Patients; Pharmacist Intervention
Keywords: polypharmacy patients; pharmacist intervention; health-related quality of life

STUDY DESIGN:
Intervention Model Description: RCT of The intervention and control groups will both have access to their physician as usual. At the medical clinic level the intervention group will receive the pharmacist intervention and other medical clinics will act as control groups. At patient level the intervention group will receive the pharmacist intervention and the control group are asked to evaluate the current treatment option.
Who Masked: Participant, Care Provider
Masking Description: The medical clinics and polypharmacy patients are blinded from the randomisation process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group - Medical clinics (Experimental): Medical clinics receiving the pharmacist intervention described in the intervention group for patient level
  Interventions: Other: Systematic pharmacist intervention
- Control group - medical clinics (No Intervention): All medical clinics that are enrolled in the trial will eventually receive the intervention at some point. As some medical clinics act as the control group to being with.
- Intervention group - patient level (Experimental): The intervention consists of two subgroups: Intervention pharmacist and intervention proposals. As the pharmacist conducts medication reviews of the polypharmacy patients in the medical clinic they can make a note to the physician about fx a specific medication the physician needs to pay attention to. These polypharmacy patients are enrolled in the group intervention proposals and are asked to complete questionaries at baseline and follow-up. Ultimately, it is up to the physician to react to the note in the polypharmacy patients medical record. Therefore the pharmacist only makes a note in the journal of the patient and does nothing else.
  The group intervention pharmacist is polypharmacy patients where the pharmacist conducts a medication review and develops suggested interventions proposals for each participant
  Interventions: Other: Systematic pharmacist intervention
- Control group - patient level (No Intervention): The control group will have access to usual care and other health services within the healthcare systems. Participants randomised to the control group are invited to participate in the evaluation of the current treatment in the primary health care sector

INTERVENTIONS:
Other: Systematic pharmacist intervention — Already described in the arm group intervention group for patient level
  Arms: Intervention group - Medical clinics; Intervention group - patient level

SUMMARY:
Brief summary: The randomised controlled trial investigates the effect of a pharmacist intervention targeting polypharmacy patient at two levels medical clinics and patient level. The purpose is to gain more knowledge to patients and physicians about their medication and to see changes in the patient's medication and health-related quality of life.

DETAILED DESCRIPTION:
The main objective of the randomised controlled trial is to investigate the clinical effects of the roll-out of the systematic offer from Nord-KAP in the North Denmark Region at two different levels (medical clinic and patient-level). The primary outcome is changes in the participant's medicine from baseline to follow up and changes in healthcare usage Secondary outcomes include investigation of cost-effectiveness and changes in patients health-related quality of life.

The hypothesis is that the regional intervention delivered by the pharmacists, from Nord-KAP, can lead to a decrease in medical products compared with a control group between baseline and at 6-month follow-up.

* Will the use of a pharmacists intervention lead to a decrease in the number of polypharmacy patients in medical clinics compared to a control group of medical clinics?
* Will the use of a pharmacist intervention lead to an increase in the polypharmacy patients health-related quality of life compared to a control group?

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 5 medicinal products prescribed besides skin remedies and antibiotic
* Above 18 years
* Patients in continuous medication treatment

Exclusion Criteria:

* Terminal patients
* Patients who are not motivated to comply with the instruction of the trial
* Do not speak/or understand written Danish
* Patients lacking legal capacity
* Patients living at nursing homes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in polypharmacypatients medication | 6 months
  The primary outcome at patient level is changes in the patients medication use at baseline and 6-month follow-up defined as the amount of medicine prescribed. Measuring the amount of medicine is extracted by the pharmacist from the participants SMC.

SECONDARY OUTCOMES:
Health-related quality of life | 6 months
  HRQoL as measures of effect for the economic evaluations. HRQoL is measured by the EQ-5D-5L questionnaire and converted into quality of life which is a scale from o to 1 where 0 correspondts to death and 1 indicates perfect health
Healthcare services | 6 months months and long term follow-up
  Use of healthcare services to estimate costs for the economic evaluation. Use of health care services are measured by Danish health registers.
Healthcare services | Up to 10 years
  Use of healthcare services to estimate costs for the economic evaluation. Use of health care services are measured by Danish health registers.
Amount of medicine pr patient in each medical clinic | 6 months
  The primary outcome for the medical clinics are changes in the patients medication at baseline and at six months follow-up
Medical clinic number of polypharmacy patients | 6 months
  . A count of the total number of polypharmacy patients in each medical clinic is conducted at baseline and six months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- The quality unit for genreal practice, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to the homepage of the pharmacist intervention from the quality unit for general practice north denmark region — https://vpvp.dk/